CLINICAL TRIAL: NCT00575562
Title: Phase I Study of KRN330 Monoclonal Antibody in Patients With Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRN330-US-01
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — KRN-330

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: KRN330 — Open-label, dose-escalation study of KRN330 in patients with relapsed or refractory advanced or metastatic colorectal cancer

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of KRN330 in patients with relapsed or refractory advanced or metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically confirmed colorectal cancer that is advanced or metastatic with measurable or assessable disease.
2. Are not candidates for a surgically curative procedure.
3. Have progressed despite, are intolerant of, or are not appropriate for current therapies.

Exclusion Criteria:

1. Have an active, uncontrolled infection.
2. Have known or suspected cerebral metastasis.
3. Have had a myocardial infarction (MI) or cerebrovascular accident (CVA) within the last 6 months; or meet the criteria for AHA class III or IV congestive heart failure (CHF).
4. Have any significant concurrent disease or illness that would interfere with the interpretation of study results.
5. Pregnant or breastfeeding women and male or female patients who do not agree to use effective contraceptive method(s) during the study.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to assess the safety and tolerability of KRN330 in patients with relapsed or refractory advanced or metastatic colorectal cancer. | For up to12 weeks

SECONDARY OUTCOMES:
The secondary objectives are to determine the degree of immunogenicity, gain information on the pharmacokinetic profile, assess the anti-tumor effects of KRN330 and determine the maximum tolerated dose (MTD). | For up to12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Berlin, M.D., Principal Investigator — Ingram Professor of Cancer Research, Vanderbilt University; Howard A Burris, III, M.D., Principal Investigator — SCRI Development Innovations, LLC
Locations (2):
- United States (2):
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee